CLINICAL TRIAL: NCT02603458
Title: A Placebo-controlled Two-dose Trial of NRX-1074 Early in the Course of Schizophrenia
Brief Title: NRX-1074 in Early Course Schizophrenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn by the sponsor.
Sponsor: NYU Langone Health (Other)
Collaborators: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S14-01975
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Naurex; Intravenous Treatment; NRX-1074
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Group of enrolled subjects receiving two infusions of intravenous placebo (5% glucose solution)
  Interventions: Drug: Placebo
- NRX-1074 Dose Group (Experimental): Group of enrolled subjects receiving two infusions of intravenous NRX-1074 (10 mg)
  Interventions: Drug: NRX-1074

INTERVENTIONS:
Drug: NRX-1074 — Participants will receive two IV NRX-1074 infusions 1 week apart, each lasting 1 minute.
  Arms: NRX-1074 Dose Group
Drug: Placebo — Patients will receive two IV placebo infusions 1 week apart, each lasting 1 minute.
  Other Names: Sugar IV solution
  Arms: Placebo

SUMMARY:
This study seeks to examine the effectiveness of NRX-1074 in the treatment of negative symptoms and cognition in schizophrenia compared to other agents at the glycine site which have demonstrated inconsistent results for negative symptoms. In addition to testing efficacy, we will examine the time course of response of symptoms as well as any effects on memory consolidation.

DETAILED DESCRIPTION:
Investigators propose to conduct a 4-week, randomized, double-blind, placebo-controlled trial in which NRX-1074 will be intravenously administered twice. Subjects will be 62 stable patients ages 18-50 within five years of onset of schizophrenia, treated with any antipsychotic except clozapine at an adequate, stable dose for at least 8 weeks. This study will be conducted by the Schizophrenia Program of the NYU Langone Medical Center and at the Psychiatry Outpatient Clinic of Bellevue Hospital located in New York, NY.

Upon signing consent, patients will undergo screening procedures to assess eligibility. A diagnosis of schizophrenia or schizophreniform disorder will be determined by the Structured Clinical Interview for DSM IV (SCID) completed by a research clinician using all available clinical data and will be confirmed by consensus diagnosis. A comprehensive medical review and physical exam, including routine laboratory tests, will be completed to identify unstable medical illness. A urine toxicology screen and, in females, a pregnancy test will also be performed. A research assistant will complete the Logical Memory Test portion of the Weschler Memory Scale-III (WMS-III).

Subjects who meet study eligibility criteria will complete the baseline visit which will include a one minute infusion of NRX-1074 and the following clinical assessments: Brief Psychiatric Rating Scale (BPRS), Clinical Assessment Interview for Negative Symptoms (CAINS), Calgary Depression Scale for Schizophrenia (CDSS), InterSePT Scale for Suicidal Thinking (ISST), Clinical Global Impression (CGI), and Systematic Assessment for Treatment Emergent Events (SAFTEE). The BPRS, SAFTEE, and ISST will be conducted twice, both before and after the infusion. The remaining assessments will be conducted before the infusion. A cognitive assessment, the Logical Memory Test of the WMS-III, will also be conducted after the infusion.

Patients will return for a visit one day after their baseline infusion, where the BPRS, ISST, CGI, and Logical Memory Test will be conducted. Their next visit will be one week later, where they receive their second NRX-1074 infusion, and will be similar in format to the first baseline infusion with the exception of CAINS and CDSS. One day after the second infusion, patients will be administered the BPRS, CAINS, CDSS, ISST, CGI, and MATRICS Consensus Cognitive Battery (MCCB). Patients will then return weekly for three weeks until Day 28.

The BPRS and ISST will be conducted during the Baseline, Day 1, Day 7, Day 8, Day 14, Day 21, and Day 28 visits. The CGI will be administered during Baseline, Day 1, Day 7, Day 8, Day 14, and Day 28. The CAINS and CDSS will be administered at Baseline, Day 8, Day 14, and Day 28. The SAFTEE will be conducted on Baseline, Day 7, Day 14, Day 21, and Day 28. The Logical Memory Test will be administered during Screening Visit 1, Screening Visit 2, Baseline, and Day 1. The MATRICS will be conducted on Day 8 and Day 28.

The primary outcome measure is the change in BPRS total score from Baseline to 24 hours post infusion on Day 8. Secondary outcome measures include the positive and negative symptom subscales on the BPRS, the CAINS total score, the composite score on the MATRICS 24 hours after the second infusion and the Logical Memory Test compared to placebo one hour after the first infusion (Baseline).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Diagnosis of Schizophrenia, Schizophreniform, or schizoaffective disorder as per DSM-V criteria
* Within five years of onset of illness
* Treated with any antipsychotic agent except clozapine at an adequate, stable dose for at least 8 weeks.
* A score of at least 4 (moderate) on at least one BPRS negative symptom item.

Exclusion Criteria:

* Serious or unstable medical illness
* Pregnant or nursing
* Abuse of substances except nicotine in the previous 6 weeks (excluding cannabis use)
* Positive urine toxicology at screening
* Experiencing serious suicidal or homicidal ideation within six months
* Treatment with clozapine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) total score | Day 8

SECONDARY OUTCOMES:
Change in total score of Brief Psychiatric Rating Scale (BPRS) from baseline to Day 28 | Baseline to Day 28
  At each time point (Day 1, Day 7, Day 8, Day 14, Day 21), contrasts between GLYX-13 and placebo will be obtained. The overall contrasts for combined GLYX-13 dose group against placebo were also estimated and tested at each time point.
Change in total score of Clinical Assessment Interview for Negative Symptoms (CAINS) from baseline to day 28 | Baseline to Day 28
  At each time point (Day 8, Day 14), contrasts between GLYX-13 and placebo will be obtained. The overall contrasts for combined GLYX-13 dose group against placebo were also estimated and tested at each time point.
Total score of MATRICS Consensus Cognitive Battery | Day 8
Total score of MATRICS Consensus Cognitive Battery | Day 28
Logical Memory Test of the Wechsler Memory Scale III | At Screening
Logical Memory Test of the Wechsler Memory Scale III | Baseline
Logical Memory Test of the Wechsler Memory Scale III | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Goff, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York University Langone Medical Center/ Bellevue Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided
The study has been withdrawn by the sponsor, so the plan to share data has not been discussed and is undecided.